CLINICAL TRIAL: NCT00247143
Title: Prospective Open Label Non-Comparative Study of the Safety, Efficacy and Tolerability of High Dose Ritonavir/Lopinavir Liquid in Salvage Therapy for PI Resistant HIV & a PK Equivalence Sub-Study of High Dose Ritonavir/Lopinavir Capsules
Brief Title: High Dose Ritonavir/Lopinavir Liquid Formulation in Salvage Therapy for Protease Inhibitor Resistant HIV Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lampiris, Harry W., M.D. (Individual)
Collaborators: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HWL-001
Record Dates: First submitted 2005-10-28; First posted 2005-11-01 (Estimated); Last update posted 2006-09-20 (Estimated); Status verified 2006-09

CONDITIONS: HIV; AIDS
Keywords: Protease Inhibitor; Antiretroviral Agents; Treatment Experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — lopinavir-ritonavir drug combination; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Kaletra (drug)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of higher doses of lopinavir/ritonavir, in combination with other anti-HIV medications when administered as either the capsule or liquid formulations, among patients who have not had full viral suppression despite treatment with 3 classes of HIV medications, and at least 2 prior courses of treatment with HIV protease inhibitors. In addition, pharmacokinetics of the active agents, lopinavir and ritonavir will be measured following administration of both the liquid and capsule formulations and compared.

DETAILED DESCRIPTION:
This study is a safety, efficacy, and tolerability study of high dose kaletra in patients who have failed multiple antiretroviral regimens, including prior treatment with 3 classes of antiretroviral drugs (nucleoside/nucleotide analogues, non-nucleoside analogues, and at least one protease inhibitor based ARV regimen), in conjunction with optimized background therapy. Patients will initially be treated with high dose kaletra capsules and optimized background therapy for 4 weeks and then switched to equivalent doses of high dose kaletra liquid formulation for a total duration of therapy of 24 weeks. The primary endpoint of the study will be the average HIV RNA change from baseline through 24 weeks (HIV RNA AACUMB). Secondary endpoints will include the proportion achieving HIV RNA < 50 and HIV RNA < 400 copies/mL at 24 weeks. Changes in CD4 from baseline, change in LPV fold change in phenotypic resistance testing, changes in fasting metabolic parameters, assessment of safety at week 24 based upon hematology, chemistry, liver function, lipid levels, proportion of patients reporting adverse events and proportion of patients with SAEs, and demonstration of bioequivalence by 12 hour pharmacokinetic measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to trial participation.
2. HIV-1 infected males or females at least 18 years of age.
3. Weight > 60 kg and < 100 kg
4. Acceptable laboratory screening values as defined in the exclusion criteria.
5. Three class ARV experienced, including current PI regimen for at least 12 weeks, at least one other PI based regimen for at least 12 weeks, treatment with at least one NNRTI and with at least 2 nucleoside agents.
6. Screening Virologic Phenotype demonstrating lopinavir phenotypic fold resistance between 10 and 80 (if patients have had Virologic Phenotype within 8 weeks of study screening this may be used as the qualifying lopinavir phenotypic fold resistance).
7. HIV-1 viral load 1000 copies/mL at screening.
8. Acceptable screening laboratory values that indicate adequate baseline organ function. Laboratory values are considered to be acceptable if the following apply:

   * Total Cholesterol ≤ DAIDS Grade 3
   * Total Triglycerides ≤ DAIDS Grade 3
   * ALT and AST ≤DAIDS Grade 3).
   * Any Grade GGT is acceptable.
   * Any Grade CK is acceptable as long as there is no concurrent myopathy.
   * All other laboratory test values ≤DAIDS Grade 2.
9. Willingness to discontinue treatment with NNRTIs throughout 48 weeks of study participation (prior or current treatment with enfuvirtide is permitted).
10. Acceptable medical history, as assessed by the investigator, with an unremarkable chest X-ray and ECG within 1 year of study participation.
11. Willingness to abstain from ingesting substances during the study which may alter plasma study drug levels by interaction with the cytochrome P450 system (these are listed in the informed consent under the risks of lopinavir/ritonavir).
12. A prior AIDS-defining event is acceptable as long as it has resolved or the patient has been on stable therapy for at least 12 weeks.

Exclusion Criteria:

1. ARV medication naïve.
2. Patients on recent drug holiday, defined as off ARV medications for at least 7 consecutive days within the last 28 days
3. Female patients of child-bearing potential who:

   * have a positive serum pregnancy test at screening or during the study,
   * are breast feeding,
   * are planning to become pregnant,
   * are not willing to a use barrier method of contraception, or
   * require ethinyl estradiol administration.
4. Prior high-dose LPV/RTV therapy (higher than recommended doses in package insert).
5. Active diarrhea not controlled with antidiarrheal medications (not to exceed 3 bowel movements/day), malabsorption, or GI intolerance to lopinavir/ritonavir
6. Use of investigational medications within 30 days before study entry or during the trial.
7. Are receiving medications that are contraindicated with, or result in significant drug-drug interactions, with LPV and/or RTV (including, but not limited to triazolam, astemizole, ergot medications, cisapride, midazolam, bepridils, or rifampin).
8. Use of immunomodulatory drugs within 30 days before study entry or during the trial (e.g. interferon, cyclosporin, hydroxyurea, interleukin 2).
9. Active malignancy requiring chemotherapy or radiation.
10. Inability to adhere to the requirements of the protocol, including active substance abuse as assessed by the investigator.
11. In the opinion of the investigator, likely survival of less than 6 months because of underlying disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-10

PRIMARY OUTCOMES:
To evaluate the safety and efficacy of high dose kaletra liquid and capsules in the treatment of highly antiretroviral experienced, protease inhibitor resistant HIV disease.

SECONDARY OUTCOMES:
To compare traditional pharmacokinetic measures of the two formulations (kaletra liquid and kaletra capsules) in a subset of the patients included in the primary analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Harry W. Lampiris, M.D., Principal Investigator — San Francisco Veterans Affairs Medical Center
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States